CLINICAL TRIAL: NCT04750499
Title: Treatment of Complex Perianal Fistulas, in Patients Without Crohn's Disease, by Endorectal Advancement Flap Associated With Injection of Autologous and Micro-fragmented Adipose Tissue
Brief Title: Treatment of Perianal Fistulas by Endorectal Advancement Flap Associated With Adipose Tissue Injection
Acronym: Fistula_CM1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fistula_CM1
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Anal Fistula
Keywords: Complex Anal Fistula; Mesenchymal Stem Cells; Microfragmented adipose tissue; Regenerative Medicine
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients with complex anal fistulas, non related to Crohn's disease.
  Interventions: Procedure: Adipose tissue injection associated with endorectal advancement flap.

INTERVENTIONS:
Procedure: Adipose tissue injection associated with endorectal advancement flap. — Injection of adipose tissue will be associated with endorectal advancement flap technique. In blind fistulas and special cases, in which the flap is not indicated, alternative techniques will be used. In all cases, autologous, micro-fragmented and minimally manipulated adipose tissue, obtained with a standardized procedure, previously validated and authorized, will be injected. This procedure uses the "Lipogems ®" device (Lipogems International SpA, Milan, Italy), with which a well-characterized adipose tissue is obtained with the maximum safety guarantees.

SUMMARY:
The study aims to evaluate effectiveness of the association of endorectal advancement flap technique with local injection of autologous and micro-fragmented adipose tissue, obtained with the Lipogems® system, in patients with complex Perianal Fistulas not related to Crohn's Disease.

DETAILED DESCRIPTION:
Treatment of anal fistula pursues permanent healing and preservation of anal continence, not always easy goals in complex anal fistulas.

In patients with Crohn's disease, simple surgery (ligation of the path and suturing of the internal orifice) associated with injections of stem cells derived from autologous or allogeneic adipose tissue has been shown to cure up to 70%. of the cases. Similar results have been obtained in small series of patients with fistulas of cryptoglandular origin and also in rectourethral and rectovaginal fistulas of other etiologies. Unfortunately, this treatment is time consuming and extremely expensive.

Fresh adipose tissue is an alternative source of mesenchymal stem cells (MSC) with regenerative capabilities, immunomodulatory angiogenic and anti-inflammatory effects. The injection of fresh adipose tissue, obtained by liposuction from the same patient, is currently a therapeutic alternative used in regenerative medicine, plastic and orthopedic surgery indications, as well in other fields. Beneficial effects of fresh adipose tissue on anus fistulas and fecal incontinence have also been reported.

The aim of the present study is to evaluate the effectiveness of the injection of autologous, microfragmented and minimally manipulated adipose tissue, associated with a surgical technique that obtains by itself up to 70% cure in order to add the benefits of surgery with those in regenerative medicine hoping that the beneficial effects of MSC will aid in the healing and repair process.

A prospective study is proposed in 12 patients with non-Crohn's-related complex anals fistulas. Whenever possible, the endorectal advancement flap technique will be applied; in blind fistulas and special cases, in which the flap is not indicated, alternative techniques will be used. In all cases, autologous, micro-fragmented and minimally manipulated adipose tissue, obtained with a standardized procedure, previously validated and authorized, will be injected. This procedure uses the "Lipogems ®" device (Lipogems International SpA, Milan, Italy), with which a well-characterized adipose tissue is obtained with the maximum safety guarantees.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, aged over 18 years old.
* Diagnosis, confirmed by standard methods (magnetic resonance and/or trans-anal ultrasound), of complex fistula (trans-sphincteric unsuitable for treatment lay-open).
* Seton placed at least 4-6 weeks previously.
* No limitations to a periodic follow-up lasting for a total of 12 months
* Informed consent form signed.

Exclusion Criteria:

* Active septic process.
* Patients unable to follow the pathway required by the protocol.
* Pregnant women.
* Failure to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Healing rate | 1 year
  Fistula tract closing by clinically assessment and confirmation by pelvic MRI if necessary.

SECONDARY OUTCOMES:
Incontinence rate | 1 year
  Presence of Fecal Incontinence Measured by the Wexner score instrument, The scoring of the instrument ranges from 0 (no incontinence) to 20 (complete incontinence).
Treatment related adverse events | 1 year
  Reported adverse events designated as related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Guillaumes, MD PhD, Principal Investigator — Hospital Clinic of Barcelona; Nils Jimmy Hidalgo, MD, Principal Investigator — Hospital Clinic of Barcelona; Irene Bachero, MD, Principal Investigator — Hospital Clinbic. Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naldini G, Sturiale A, Fabiani B, Giani I, Menconi C. Micro-fragmented adipose tissue injection for the treatment of complex anal fistula: a pilot study accessing safety and feasibility. Tech Coloproctol. 2018 Feb;22(2):107-113. doi: 10.1007/s10151-018-1755-8. Epub 2018 Feb 16. PMID 29453515
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Herreros MD, Garcia-Arranz M, Guadalajara H, De-La-Quintana P, Garcia-Olmo D; FATT Collaborative Group. Autologous expanded adipose-derived stem cells for the treatment of complex cryptoglandular perianal fistulas: a phase III randomized clinical trial (FATT 1: fistula Advanced Therapy Trial 1) and long-term evaluation. Dis Colon Rectum. 2012 Jul;55(7):762-72. doi: 10.1097/DCR.0b013e318255364a. PMID 22706128
- [Background] Bianchi F, Maioli M, Leonardi E, Olivi E, Pasquinelli G, Valente S, Mendez AJ, Ricordi C, Raffaini M, Tremolada C, Ventura C. A new nonenzymatic method and device to obtain a fat tissue derivative highly enriched in pericyte-like elements by mild mechanical forces from human lipoaspirates. Cell Transplant. 2013;22(11):2063-77. doi: 10.3727/096368912X657855. Epub 2012 Oct 8. PMID 23051701
- [Background] Tremolada C, Ricordi C, Caplan AI, Ventura C. Mesenchymal Stem Cells in Lipogems, a Reverse Story: from Clinical Practice to Basic Science. Methods Mol Biol. 2016;1416:109-22. doi: 10.1007/978-1-4939-3584-0_6. PMID 27236668
- [Derived] Guillaumes S, Hidalgo NJ, Bachero I, Pena R, Nogueira ST, Ardid J, Pera M. Efficacy of injection of autologous adipose tissue in the treatment of patients with complex and recurrent fistula-in-ano of cryptoglandular origin. Tech Coloproctol. 2024 Jul 9;28(1):81. doi: 10.1007/s10151-024-02963-x. PMID 38980511